CLINICAL TRIAL: NCT07193862
Title: Pilot Study of an Implantable Microdevice for In Situ Evaluation of Drug Response in Patients With Colorectal Liver Metastasis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0004
Record Dates: First submitted 2025-09-03; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Doxorubicin; Folfox protocol; balstilimab; Bevacizumab; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): Subjects will have the device placed loaded with chemotherapeutic agents.
  Interventions: Combination Product: Doxorubicin, FOLFOX, Botensilimab, Balstilimab, Bevacizumab, FOLFIRI, FOLFIRINOX, AGEN2373

INTERVENTIONS:
Combination Product: Doxorubicin, FOLFOX, Botensilimab, Balstilimab, Bevacizumab, FOLFIRI, FOLFIRINOX, AGEN2373 — Patients with diagnosed liver metastasis from a colorectal primary deemed resectable. The study intervention will be limited to the percutaneous placement of up to 2 IMDs per lesion with a maximum of 4 devices total, with the subsequent en bloc resection of the tumor plus IMD within 3 (+2) days after placement. The microdevices will remain in the tumor for a minimum of a 2-day incubation period, although ideally for 3 days.
  The IMD is a small cylindrical device approximately 750 um in diameter and 5 mm in length (Figure 2), housing up to 21 reservoirs. It is made of PEEK, biocompatible material used in other implantable constructs, including joint replacements. 11-13 Drugs are solubilized with poly-ethylene glycol (PEG) and loaded into the individual reservoirs. The drug diffusion has been mapped extensively to ensure that the weight of PEG is selected such that drug diffusion is limited and will not mix or interfere with another drug.

SUMMARY:
Microdevices have been used to ascertain in vivo drug response, which can lead to improved cancer treatment delivery; however, they have not been evaluated for liver tumors. This is a prospective, phase 1 safety study of percutaneous placement and surgical retrieval of a microdevice in patients with liver metastasis from colorectal cancer. The device will be implanted percutaneously 3-5 days prior to scheduled resection of colorectal liver metastasis (CLM) and then removed en bloc with the tumor. Patients will be monitored to ensure that the device's placement and retrieval does not result in increased complication rates within 14 days of surgery. To assess feasibility, the tissue surrounding the microdevice will be analyzed to assess the diffusion of the drugs from the device into the tissue and whether the therapeutic effect of diffusing chemotherapy +/- immune-modulating drugs has an impact on the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer with suspicion of liver metastasis on imaging Liver tumor ≥2 cm on preoperative imaging via computed tomography (CT) or magnetic resonance imaging (MRI) Planned hepatectomy as part of standardized treatment plan, irrespective of study enrollment ≥18 years of age

Normal organ and marrow function, defined as follows:

* Leukocytes ≥3,000/mcL
* Absolute neutrophil count ≥1500/mcL
* Platelets ≥ 100,000/mcL
* PT≤ 14, PTT≤ 38, INR ≤ 1.
* Creatinine within normal institutional limits OR clearance ≥60mL/min/1.73m2 Feasibility of microdevice implantation based on clinical history as well as extent and anatomical location of the CLM tumor as evaluated by the operating surgical oncologist and interventional radiologist on baseline imaging The effects of the microdevice on a developing human fetus are unknown. For this reason and because the therapeutic agents used in this trial are known to be teratogenic, women of childbearing age must agree to have a negative serum pregnancy test within 48 hours of their operation Ability to understand and willingness to sign informed consent for both the surgical resection and the proposed research study prior to any procedures

Males and females of childbearing potential must agree to use effective contraception starting before the first day of treatment and continuing for at least 3 months (men) or 6 months (women) after implantation of the microdevice. Additionally, due to the unknown but potential risks of nursing infants secondary to the treatment of the mother with the chemotherapeutic agents of the study, mothers must agree to discontinue breastfeeding for a total of 14 days after the insertion of the microdevice.

Exclusion Criteria:

Tumor location not amenable to device placement Pregnancy at the time of enrollment or operation due to the known teratogenicity of the medications involved.

Prior or concurrent second primary malignancy whose natural history or treatment has the potential to interfere with the safety or primary endpoint efficacy assessment of the CLM Extra-hepatic disease or unresectable liver metastasis on baseline imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) associated with Microdevice placement and retrieval | 12 months
  To evaluate the safety of microdevice placement and retrieval based on assessment of adverse events.
  AEs will be defined using Common Terminology Criteria for AEs (CTCAE) v5.0
  Any device resulting in either of the following will be considered a failure from a safety standpoint:
  any listed SAE two or more grade 3-4 AEs directly associated with the device or its placement
  Significant delay in the standard hepatic resection of more than 14 days due to device-related complications
  Safety will be evaluated on a per-patient level, where an event is defined as any "failure" observed among all devices.
  This is a phase 1 pilot safety trial that must only demonstrate the ability to perform this procedure without undue risk

CONTACTS AND LOCATIONS:
Locations (1):
- RJ Zuckerberg, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No